CLINICAL TRIAL: NCT04053907
Title: P. Falciparum Infection Dynamics and Transmission to Inform Elimination
Acronym: INDIE-1b
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); National Malaria Control Programme, The Gambia (Other Government); Radboud University Medical Center (Other); University of California, San Francisco (Other); Institute for Disease Modeling (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16642; OPP1173572 (Other Grant/Funding Number: Bill and Melinda Gates Foundation (BMGF))
Record Dates: First submitted 2019-07-29; First posted 2019-08-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Malaria
Keywords: falciparum; gametocyte; elimination; anopheles; transmission; diagnostic
MeSH Terms: conditions — Malaria; Disease | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CCM:Standard of Care (No Intervention): Community Case Management (CCM), with passively monitored malaria incidence by community health workers using standard RDTs and artemisinin-based combination therapy (ACT), artemether-lumefantrine (AL) according to national guidelines.
- CCM plus weekly fever screening and treatment (Experimental): CCM plus active case detection (ACD) by fever screening and treatment if positive. Trained village health workers (VHW) recruited for this study will carry out weekly visits of all residents and screen for fever using research-grade thermometers. A standard RDT will be performed in all individuals with a body temperature ≥37.5°C or with reported fever in the last 24 hours. RDT positive individuals will be treated with AL according to national guidelines.
  Interventions: Other: Community Case Management; Other: Weekly fever screening and treatment
- CCM plus MSAT (Experimental): CCM plus monthly screening for malaria infection and treatment of positive individuals, regardless of symptoms. Screening will be performed by research staff and timed to ensure a gap of 25-35 days between screening rounds; Positive individuals will be treated with AL, according to national guidelines.
  Interventions: Other: Community Case Management; Other: Monthly malaria screening
- CCM plus dry season MDA (Experimental): CCM plus plus 3 monthly rounds of MDA with a long-acting ACT (dihydroartemisinin-piperaquine, DP) starting in the dry season (April, May, June) (tablets of 320/40mg and 160/20mg piperaquine/ dihydroartemisinin per tablet. Administration of a full course of DP will be done as per manufacturer's guidelines once daily for 3 days and according to body weight).
  Interventions: Other: Community Case Management; Other: MDA

INTERVENTIONS:
Other: Community Case Management — Community Case Management (CCM), consisting of community health workers able to diagnose malaria by standard RDTs and treating positive individuals with artemether-lumefantrine (AL), according to national guidelines.
  Arms: CCM plus MSAT; CCM plus dry season MDA; CCM plus weekly fever screening and treatment
Other: Weekly fever screening and treatment — Consists of weekly visits by trained VHW who will screen for fever by taking the axillary temperature. If the body temperature is ≥37.5°C, a standard RDT will be performed and, if positive, the individual will be treated with AL, according to national guidelines.
  Arms: CCM plus weekly fever screening and treatment
Other: Monthly malaria screening — CCM plus monthly screening of the whole population with high sensitive RDT (HS-RDT); positive individuals will be treated with AL regardless of symptoms (MSAT).
  Arms: CCM plus MSAT
Other: MDA — CCM plus 3 monthly rounds of MDA with dihydroartemisinin-piperaquine (DP) starting during the dry season, before the malaria transmission season starts.
  Arms: CCM plus dry season MDA

SUMMARY:
In the current study, three experimental approaches aiming at reducing malaria transmission will be tested. The study will cover two transmission season (2019 and 2020) and the interventions will vary by season. More specifically, in the 2019 transmission season (June-December) (Year 1), community case management of malaria (CCM) will be implemented in all eight villages as improved standard of care; in the 2020 transmission season (Year 2), the eight study villages will be divided into 4 study arms. CCM will continue in all villages; two villages will continue with CCM only (Arm 1, control); the three other pairs of villages will receive active fever screening and treatment (Arm 2); monthly mass screening and treatment (MSAT) (Arm 3); and mass drug administration (MDA) during the last 3 months of the dry season (April-June) (Arm 4). For MDA, the whole population (except for those not fulfilling the entry criteria) will be treated with a full course of dihydroartemisinin-piperaquine (DP) (320/40mg and 160/20mg piperaquine/ dihydroartemisinin per tablet) per manufacturer's guidelines (once daily for 3 days and according to body weight). The MDA treatment will be repeated 3 times at monthly intervals.

DETAILED DESCRIPTION:
In the current study, the investigators will first improve access to care in all villages by implementing community-based clinical case management (CCM) (year 1). In this year, the investigators will quantify gametocyte carriage and transmission from clinical cases passively recruited by CCM, and gametocyte carriage and transmission from asymptomatic infections detected in community surveys. These data will support the interpretation of the main study outcomes in year 2 when the investigators will directly compare the effect of CCM on the human reservoir of infection as compared to three different approaches, namely i) active fever screening and treatment that should detect symptomatic infections for early treatment; ii) Mass Screening and Treatment (MSAT) that will systematically screen, using point-of-care diagnostics, the whole population, with infected individuals immediately treated; and iii) mass drug administration (MDA) that will treat the whole population with a full course of an antimalarial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Resident in the village.
2. Willingness to participate in repeated assessments of health and infection status and to donate a maximum of 30 mL (milliliter) of blood (children <5 years of age), 37 mL (milliliter) of blood (children <10 years of age) or 52 mL (milliliter) of blood (older individuals) during an 18-month period.

Exclusion Criteria:

1. Any chronic illness that would affect study participation.
2. Pre-existing severe chronic health conditions
3. History of intolerance to artemether-lumefantrine.
4. Participants < 6months old and pregnant women in the first trimester (only for Arm with MDA-DP treatment).
5. Hypersensitivity to DP (only for Arm with MDA-DP treatment).
6. Taking drugs that influence cardiac function or prolong QTcorrected interval (only for Arm with MDA-DP treatment).

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Parasite prevalence by molecular detection at the end of study (cross-sectional survey). | 16 weeks
  The primary outcome measure is parasite prevalence in the cross-sectional survey conducted at the end of the transmission season of year 2.
Parasite density by molecular detection at the end of study (cross-sectional survey). | 16 weeks
  The primary outcome measure is parasite density (parasite/µL) in the cross-sectional survey conducted at the end of the transmission season of year 2.

SECONDARY OUTCOMES:
Gametocyte prevalence by molecular methods at the end of study (cross-sectional survey). | 16 weeks
  Gametocyte prevalence in quantitative polymerase chain reaction (qPCR) detected infections is assessed by molecular methods and compared between arms.
Gametocyte density by molecular methods at the end of study (cross-sectional survey). | 16 weeks
  Gametocyte density (gametocytes/µL) in qPCR detected infections is assessed by molecular methods and compared between arms.
Gametocyte prevalence of male and female gametocytes by molecular methods among P. falciparum infections at all study visits. | Throughout study, an average of 18 months
  Gametocyte prevalence of male and female gametocytes will be assessed by molecular methods and compared between study arms.
Gametocyte density of male and female gametocytes by molecular methods among P. falciparum infections at all study visits. | Throughout study, an average of 18 months
  Gametocyte density of male and female gametocytes will be assessed by molecular methods and compared between study arms.
Incidence of malaria infections | Throughout study, an average of 18 months
  Regular visits by weekly active case detection and monthly screening will result in the identification of malaria infections that are not detected during CCM. Number of infections detected in each arm will be quantified and compared between arms.
Infectivity of P. falciparum infections to mosquitoes | Throughout study, an average of 18 months
  For a selection of infections, infectiousness to mosquitoes is assessed by membrane feeding assays.

OTHER OUTCOMES:
The detectability of infections by highly-sensitive rapid diagnostic tests related to histidine rich protein-2 (HRP2) concentrations. | Throughout study, an average of 18 months
  For a selection of samples, the detectability of infections is assessed by highly sensitive rapid diagnostic tests related to histidine rich protein-2 (HRP2) concentrations.
The detectability of infections by highly-sensitive rapid diagnostic tests related to duration of infection. | Throughout study, an average of 18 months
  For a selection of samples, the detectability of infections is assessed by highly sensitive rapid diagnostic test and related to duration of infection.
The detectability of infections by rapid diagnostic tests related to duration of infection. | Throughout study, an average of 18 months
  For a selection of samples, the detectability of infections is assessed by conventional rapid diagnostic tests and related to duration of infection.
The detectability of infections by highly-sensitive rapid diagnostic tests related to parasite density by molecular diagnostics. | Throughout study, an average of 18 months
  The detectability of infections is assessed by highly sensitive rapid diagnostic test and related to parasite density by molecular diagnostics.
The detectability of infections by rapid diagnostic tests related to parasite density by molecular diagnostics. | Throughout study, an average of 18 months
  For a selection of samples, the detectability of infections is assessed by conventional rapid diagnostic test and related to parasite density by molecular diagnostics.
The relationship between the proportion of infected mosquitoes (Direct Membrane Feeding Assay) and gametocyte density. | Throughout study, an average of 18 months
  Gametocyte density will be assessed by molecular methods and associated with infectivity mosquitoes.
The relationship between the proportion of infected mosquitoes (Direct Membrane Feeding Assay) and gametocyte sex-ratio. | Throughout study, an average of 18 months
  Sex-ratio gametocytemia of P. falciparum will be assessed by molecular methods and associated with infectivity in mosquitoes.
The effect of infection characteristics (clonal parasite infection) on the transmissibility of infections to mosquitoes. | Throughout study, an average of 18 months
  To determine the impact of duration and complexity of malaria infections on the transmissibility of infections to mosquitoes
Gametocyte sex-ratio on the transmissibility of infections to mosquitoes. | Throughout study, an average of 18 months
  To determine the impact of gametocyte sex-ratio on the transmissibility of infections to mosquitoes
The impact of human haemoglobinopathies on the transmissibility of infections to mosquitoes. | Throughout study, an average of 18 months
  To determine the impact of red blood cell haemoglobinopathies and haemoglobin concentration on the transmissibility of infections to mosquitoes.
Mean fluorescence intensity (MFI) to inflammatory markers and naturally acquired antibody responses to gametocyte antigens on the transmissibility of infections to mosquitoes. | Throughout study, an average of 18 months
  To determine the impact of inflammatory markers and naturally acquired antibody responses to gametocyte antigens and other host characteristics on the transmissibility of infections to mosquitoes.
Relationship between total parasite density (parasite/µL) and gametocyte density (gametocytes/µL) | Throughout study, an average of 18 months
  To assess the relationship between asexual parasite density and gametocyte density in P. falciparum infections
Malaria transmission potential based on measured gametocyte densities (gametocytes/µL). | Throughout study, an average of 18 months
  To determine malaria transmission potential of infections based on the gametocyte density
Number of acquired parasite clones based on genotyping. | Throughout study, an average of 18 months
  Under this outcome, we aim to examine the complexity of P. falciparum infection by measuring the number of clones present in infections
Number of days that P. falciparum infections last in the dry season. | Up to 6 months
  To evaluate the duration of P. falciparum carriage during the dry season, routine follow-up will be performed.
Mosquito exposure monitored by monthly CDC-light traps (CDC-LT) and Human landing catches (HLC) mosquito collections | Throughout study, an average of 18 months
  For the quantification of the mosquito exposure, indoor and outdoor mosquito collections will be performed monthly during transmission and dry season.
Mean fluorescence intensity (MFI) antibody responses to mosquito saliva proteins during high and low transmission season. | Throughout study, an average of 18 months
  To determine the exposure to Anopheles bites with serological markers of malaria infection.
Number of infections in community surveys that can be linked to a symptomatic or asymptomatic parent infection. | Throughout study, an average of 18 months
  This outcome allow bridging mosquito feeding studies with actual transmission events in communities and at the same time quantify the relevance of infections associated with movement.
Number of human host from mosquito blood meal source. | Up to 12 months
  To quantify the transmission potential of individuals by identification of human blood source by molecular typing.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Drakeley, PhD, Principal Investigator — London School Hygiene and Tropical medicine; Umberto D'Alessandro, PhD, MD, Principal Investigator — MRC Unit The Gambia @ LSHTM; Teun Bousema, PhD, Principal Investigator — Radboud University Medical Centre, Nijmegen, The Netherlands
Locations (1):
- Medical research Council Unit The Gambia at LSHTM, Basse Santa Su, The Gambia

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised individual participant data may be shared on a digital repository or upon reasonable request.